CLINICAL TRIAL: NCT03951207
Title: Randomized, Multicenter, Parallel, Open, Phase 4 Study to Compare the Efficacy and Safety of Rosuvastatin/Amlodipine Combination Therapy Versus Atorvastatin/Amlodipine Combination Therapy in Hypertension Patient With Dyslipidemia
Brief Title: Rosuvastatin/Amlodipine vs Atorvastatin/Amlodipine in Hypertension Patient With Dyslipidemia
Acronym: CORONA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YMC040
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2020-12

CONDITIONS: Dyslipidemias; Hypertension
MeSH Terms: conditions — Dyslipidemias; Hypertension | interventions — Amlodipine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rosuampin 10/5mg (Experimental): Rosuvastatin 10mg/Amlodipine 5mg qd for 8 weeks
  Interventions: Drug: Rosuampin 10/5mg
- Rosuampin 20/5mg (Experimental): Rosuvastatin 20mg/Amlodipine 5mg qd for 8 weeks
  Interventions: Drug: Rosuampin 20/5mg
- Amlodipine/Atorvastatin 5/20mg (Active Comparator): Atorvastatin 20mg/Amlodipine 5mg qd for 8 weeks
  Interventions: Drug: Amlodipine/Atorvastatin 5/20mg

INTERVENTIONS:
Drug: Rosuampin 10/5mg — Rosuvastatin 10mg/Amlodipine 5mg qd for 8 weeks
  Arms: Rosuampin 10/5mg
Drug: Rosuampin 20/5mg — Rosuampin 20/5mg qd for 8 weeks
  Arms: Rosuampin 20/5mg
Drug: Amlodipine/Atorvastatin 5/20mg — Amlodipine/Atorvastatin 5/20mg qd for 8 weeks
  Arms: Amlodipine/Atorvastatin 5/20mg

SUMMARY:
This study is to Compare the Efficacy and Safety of Rosuvastatin/Amlodipine Combination Therapy Versus Atorvastatin/Amlodipine Combination Therapy in Hypertension patient with Dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* Both man and woman who is over 19 years old
* Patient with dyslipidemia and hypertension
* Written informed consent

Exclusion Criteria:

* Triglyceride ≥ 400 mg/dL at screening
* Hypertensive patients who need antihypertensive medication except Amlodipine, β-blockers, RAS inhibitors
* sSBP difference is ≥20 mmHg or sDBP difference is ≥10 mmHg
* A history of rhabdomyolysis, myopathy
* Patient with hypersensitivity to Statin or Amlodipine
* Patients undergoing eGFR <30 mL/min/1.73 m2 (MDRD) at screening
* AST(Aspartate Aminotransferase) or ALT(Alanine Aminotransferase) level ≥ 3x ULN (upper limit of normal range) or active liver disease
* Creatine kinase (CK) level ≥ 5x ULN (upper limit of normal range)
* Contraindications stated in the Label of Rosuampin or Caduet
* Those participating in other clinical trials for investigational products at screening
* Patients deemed to be ineligible to participate in the trial by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Rate of change from baseline to week 8 in LDL-Cholesterol | Baseline/Week 8

SECONDARY OUTCOMES:
Rate of change from baseline to week 4 in LDL-Cholesterol | Baseline/Week 4
Proportion of subjects who reached the therapeutic goal to week 8 | Week 8
  * Group I: < 160 mg/dL, Group II: < 130 mg/dL, Group III: < 100 mg/dL
Rate of change from baseline to week 4, 8 in lipid profile(without LDL-C) | Baseline/Week 4, 8
  Total cholesterol, HDL-C, Triglyceride, Apo A-1, Apo B, Apo B/Apo A-1, Lipoprotein(a)
Rate of change from baseline to week 4, 8 in hs-CRP | Baseline/Week 4, 8
Rate of change from baseline to week 4, 8 in glucose index | Baseline/Week 4, 8
  Fasting Blood Glucose, HbA1C, HOMA-IR
Rate of change from baseline to week 4, 8 in msSBP & msDBP in both arm | Baseline/Week 4, 8
Rate of change from baseline to week 4, 8 in difference of msSBP & msDBP in both arm | Baseline/Week 4, 8
The incidence of major adverse cardiovascular and cerebrovascular events (MACCE) | Week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Daegu Catholic Univ. Medical Center, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park CM, Jung HW. Predictors of Significant High-Sensitivity C-Reactive Protein Reduction After Use of Rosuvastatin/Amlodipine and Atorvastatin/Amlodipine-Subgroup Analysis in Randomized Controlled Trials. J Clin Med. 2025 May 12;14(10):3363. doi: 10.3390/jcm14103363. PMID 40429358
- [Derived] Jung HW, Kim CY, Hong SP, Bae HJ, Choi JY, Ryu JK, Lee JB, Lee KH, Han KR, Yang DH, Park CG, Yu GW, Rhee MY, Park SJ, Hyon MS, Shin JH, Hong BK, Jin HY, Lee SY, Seol SH, Lee SR, Kim SY, Lee KJ, Cho EJ, Nam CW, Park TH, Kim U, Kim KS. Randomized, multicenter, parallel, open, phase 4 study to compare the efficacy and safety of rosuvastatin/amlodipine polypill versus atorvastatin/amlodipine polypill in hypertension patient with dyslipidemia. J Clin Hypertens (Greenwich). 2023 Sep;25(9):828-844. doi: 10.1111/jch.14715. Epub 2023 Aug 16. PMID 37584254